CLINICAL TRIAL: NCT02842918
Title: The Immediate Effects of Thoracic Spine Manipulation Versus a Sham Comparator on the Upper Limb Provocation Test and Seated Slump Test
Brief Title: The Effect of Thoracic Spine Manipulation on Peripheral Neurodynamic Mobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenandoah University (Other)
Responsible Party: Principal Investigator, Aaron Hartstein, Assistant Professor Division of Physical Therapy, Shenandoah University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ShenandoahU
Record Dates: First submitted 2016-07-19; First posted 2016-07-25 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Musculoskeletal Manipulations
Keywords: Thoracic Spine Manipulation; Neurodynamics; Sham

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spinal Manual Therapy (Active Comparator): Supine thoracic spine manipulation located between the levels of T4-T7
  Interventions: Procedure: Spinal Manual Therapy; Procedure: Spinal Range of Motion
- Spinal Range of Motion (Sham Comparator): Supine thoracic spine sham manipulation located between the levels of T4-T7; identical procedure as the active treatment intervention but without the delivery of high velocity low amplitude thrust
  Interventions: Procedure: Spinal Manual Therapy; Procedure: Spinal Range of Motion

INTERVENTIONS:
Procedure: Spinal Manual Therapy
  Other Names: Active treatment group
Procedure: Spinal Range of Motion
  Other Names: Placebo/Sham group

SUMMARY:
No studies have investigated the effects of a supine thoracic spine manipulation (TSM) on neurodynamic mobility, as compared to a sham intervention. This study aims to determine the immediate effects of TSM on the Upper Limb Provocation Test (ULPT) and Seated Slump Test (SST) compared to a sham intervention in asymptomatic subjects with neurodynamic limitations.

DETAILED DESCRIPTION:
A convenience sample will be utilized to obtain subjects. Subjects will be given a brief questionnaire to identify possible contraindications for spinal treatment techniques and exclude individuals if necessary. Subjects will be randomized into one of two groups (spinal manual therapy or spinal range of motion which will serve as the name for the placebo group) and participate in neurodynamic testing procedures of the upper extremity (Upper Limb Provocation Testing) as well as lower extremity (Seated Slump Test). Subjects who are determined to be positive for one or more limbs will receive either a thoracic spine manipulation technique (spinal manual therapy) or a thoracic spine sham manipulation technique (spinal range of motion/placebo). After application of the technique, previously positive limbs will be retested. In attempt to determine validity and believability of the sham procedure and perception of its effect, subjects will be asked if they believe their upper/lower quarter mobility will change based on the group name and after the technique is applied. Subjects will also be asked if they believed they were in the treatment or placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Upper Limb Provocation Test results with limitation of greater than 60 deg of elbow extension at the time of measurement
* Seated Slump Test results with limitation of greater than 22 deg of knee extension at the time of measurement

Exclusion Criteria:

* History of cervical or lumbar pain requiring medical intervention within the last two years, history of upper or lower extremity paresthesia/numbness, self reported bone density disorders, previous spinal cord injury, diagnosed intervertebral disc herniation, previous diagnosis of spinal stenosis or disc pathology, current pregnancy, history of circulatory or neurological disorders, history of spine and extremity fractures or dislocations in the last two years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-02; Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Upper Limb Provocation Test Range of Motion Change (measured in degrees of elbow extension) | Pre and Immediately Post Intervention
  Subjects will lie on their back with their shoulder slightly off the edge of a treatment table. The investigator will then bend the subjects neck away from the shoulder being tested and position the arm into the starting test position. The investigator will then straighten the subjects elbow until it is fully extended, or until the subject reports discomfort or an abnormal feeling in their arm. This procedure will be completed before and immediately after either the treatment intervention (manipulation) or the sham intervention is completed.
Seated Slump Test Range of Motion Change (measured in degrees of knee extension) | Pre and Immediately Post Intervention
  Subjects will sit at the edge of treatment table. Subjects will be asked to flex then neck towards their chest. The investigator will then apply a gentle force to their upper back and will ask the subject to remain in this position. The investigator will move the subjects foot upwards and straighten their leg until it is fully extended or until the subject reports discomfort or an abnormal feeling in their leg.This procedure will be completed before and immediately after either the treatment intervention (manipulation) or the sham intervention is completed.

SECONDARY OUTCOMES:
Believability of Sham - measured via questionnaire | Immediately Post Intervention (after final measurements are read and recorded)
  Subjects will be asked whether they believe they were in the active treatment group or the sham/placebo group after final measurements are taken.
Perceived effect - measured via questionnaire | Pre Intervention (immediately after initial measurements are recorded and prior to intervention)
  Subjects will be asked whether they believe their upper and/or lower quarter mobility will change based on the group name they are assigned.

CONTACTS AND LOCATIONS:
Overall Officials: Sheri A Hale, PhD, PT, ATC, Study Director — Shenandoah University
Locations (1):
- Shenandoah University, Winchester, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be available to analyze; Subject grouping will not be available to participants in attempt to control believability of the sham comparator

REFERENCES:
- [Result] Michener LA, Kardouni JR, Sousa CO, Ely JM. Validation of a sham comparator for thoracic spinal manipulation in patients with shoulder pain. Man Ther. 2015 Feb;20(1):171-5. doi: 10.1016/j.math.2014.08.008. Epub 2014 Sep 6. PMID 25261090
- [Result] Davis DS, Anderson IB, Carson MG, Elkins CL, Stuckey LB. Upper Limb Neural Tension and Seated Slump Tests: The False Positive Rate among Healthy Young Adults without Cervical or Lumbar Symptoms. J Man Manip Ther. 2008;16(3):136-41. doi: 10.1179/jmt.2008.16.3.136. PMID 19119402
- [Result] Szlezak AM, Georgilopoulos P, Bullock-Saxton JE, Steele MC. The immediate effect of unilateral lumbar Z-joint mobilisation on posterior chain neurodynamics: a randomised controlled study. Man Ther. 2011 Dec;16(6):609-13. doi: 10.1016/j.math.2011.06.004. Epub 2011 Jul 13. PMID 21742541
- [Result] Chu J, Allen DD, Pawlowsky S, Smoot B. Peripheral response to cervical or thoracic spinal manual therapy: an evidence-based review with meta analysis. J Man Manip Ther. 2014 Nov;22(4):220-9. doi: 10.1179/2042618613Y.0000000062. PMID 25395830
- [Result] Schmid A, Brunner F, Wright A, Bachmann LM. Paradigm shift in manual therapy? Evidence for a central nervous system component in the response to passive cervical joint mobilisation. Man Ther. 2008 Oct;13(5):387-96. doi: 10.1016/j.math.2007.12.007. Epub 2008 Mar 3. PMID 18316238